CLINICAL TRIAL: NCT02140502
Title: Incidence of Fluoroquinolone Resistant Bacteria in Patients Undergoing Prostate Biopsy
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); HUSLAB (Unknown)
Responsible Party: Principal Investigator, Kanerva Lahdensuo, MD, Helsinki University Central Hospital
Other Study IDs: Prostate Biopsy Infections
Record Dates: First submitted 2014-05-01; First posted 2014-05-16 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Fluoroquinolone Resistant Enteric Bacteria
Keywords: Enterobacterial Infections; Prostate cancer; Biopsy; Incidence of fluoroquinolone resistant enteric bacteria
MeSH Terms: conditions — Enterobacteriaceae Infections; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — rectal culture swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Men undergoing prostate biopsy

SUMMARY:
In this study, the investigators aim to establish the incidence of enteric fluoroquinolone resistant bacteria in a contemporary clinical cohort. This incidence will be studied by taking a rectal swab sample from all consenting patients coming in for prostate biopsies. The information gained from this study will be used to determine whether antibiotic prophylactic practices need to be updated in their clinic. The investigators aim to enroll 200 patients and patient recruitment is estimated to take place between May 2014 and August 2014. The study is estimated to end in May 2016.

DETAILED DESCRIPTION:
Due to prostate-specific antigen (PSA) screening and the aging population in many Western countries, prostate biopsies to detect prostate cancer are being taken more and more often. Prostate biopsies are also performed in the surveillance of prostate cancer. In most cases, biopsies are taken trans-rectally with ultrasound guidance. Due to the trans-rectal route, there is an inherent risk of infectious complications. These complications range from minor complications, such as bacteriuria and epididymitis, to severe complications requiring intensive care such as sepsis. The rate of these most severe complications has long been estimated at 1-2 %, but a steady rise has been observed since the beginning of the 21st century, with some centers reporting occurrence rates as high as 8%. Interestingly, the rate of other complications related to this procedure (e.g. rectal bleeding, hematuria, hematospermia, dysuria) have remained constant. Prophylactic antibiotics are routinely administered to minimize the rate of infectious complications. The most commonly used prophylactic antibiotic agents are fluoroquinolones (FQ). The observed rise in the rate of severe complications has been attributed to emerging strains of FQ-resistant bacteria. Known risk factors for harboring enteric resistant bacterial strains are recent (within three months) antibiotic use and travel to areas where these bacterial strains are known to be endemic. When a patient is known to harbor FQ-resistant enterobacteria, a different prophylactic antibiotic should be chosen. In this study, the investigators aim to prospectively establish the incidence of enteric FQ-resistant bacteria in a clinical patient cohort. This incidence will be studied by taking a rectal swab sample from all consenting patients coming in for prostate biopsies. The information gained from this study will be used mainly to determine whether antibiotic prophylactic practices need to be updated in their clinic. The investigators aim to enroll 200 patients and patient recruitment is estimated to take place between May 2014 and August 2014. The study is estimated to end in May 2016.

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion of prostate cancer or previous diagnosis of prostate cancer
* must be able to give informed consent

Exclusion Criteria:

* uncontrolled serious infection
* uncontrolled hemorrhagic disorder
* rectal swab sample not possible

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men undergoing prostate biopsy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of fluoroquinolone resistant enteric bacteria | 14 days after rectal swab
  The rectal swabs will be cultured in mediums that contain fluoroquinolones (FQ) to assess whether FQ-resistant bacterial strains emerge. The culture findings will be evaluated 14 days after obtaining the samples. The number of participants with FQ-resistant enteric bacteria is analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Antti Rannikko, MD, PhD, Principal Investigator — Helsinki University Central Hospital; Henrikki Santti, M.D., PhD, Principal Investigator — Helsinki University Central Hospital; Kanerva Lahdensuo, M.D., Principal Investigator — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Department of Urology, Meilahti Hospital, Helsinki, Uusimaa
  - Department of Urology, Peijas Hospital, Vantaa, Uusimaa

REFERENCES:
- [Derived] Kalalahti I, Huotari K, Lahdensuo K, Tarkka E, Santti H, Rannikko A, Patari-Sampo A. Rectal E. coli above ciprofloxacin ECOFF associate with infectious complications following prostate biopsy. Eur J Clin Microbiol Infect Dis. 2018 Jun;37(6):1055-1060. doi: 10.1007/s10096-018-3217-7. Epub 2018 Mar 2. PMID 29500572